CLINICAL TRIAL: NCT02183415
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses (2.5, 5, and 10 mg q.d. for 28 Days) of BI 1356 BS as Tablet in Patients With Type 2 Diabetes (Randomised, Double-blind, Placebo-controlled Within the Dose Groups)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 1356 BS as Tablet in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.3
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (4):
- BI 1356 BS, low dose (Experimental)
  Interventions: Drug: BI 1356 BS, low dose
- BI 1356 BS, medium dose (Experimental)
  Interventions: Drug: BI 1356 BS, medium dose
- BI 1356 BS, high dose (Experimental)
  Interventions: Drug: BI 1356 BS, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356 BS, low dose
  Arms: BI 1356 BS, low dose
Drug: BI 1356 BS, medium dose
  Arms: BI 1356 BS, medium dose
Drug: BI 1356 BS, high dose
  Arms: BI 1356 BS, high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 1356 BS during 4 week treatment duration

ELIGIBILITY:
Inclusion Criteria:

* Male and female postmenopausal patients with proven diagnose of type 2 diabetes mellitus treated with diet and exercise only or with one (or two) oral hypoglycaemic agents besides glitazones
* Glycosylated haemoglobin A1 (HbA1c)

  * ≤ 8.5 % at screening for patients treated with diet and exercise and/or one oral hypoglycaemic agent or
  * ≤ 8.0 % at screening for patients treated with two oral hypoglycaemic agents
* Male patients: Age ≥21 and Age ≤70 years
* Female patients: Age ≥60 and Age ≤70 years
* BMI ≥18.5 and BMI ≤35 kg/m2 (Body Mass Index)
* Caucasian ethnicity
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including Blood Pressure, Pulse Rate and Electrocardiogram) deviating from normal and of not acceptable clinical relevance
* Clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency NYHA (New York Heart Association) II-IV, known cardiovascular diseases including hypertension > 150/95mmHg, stroke and TIA (transient ischemic attack)
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes, hyperlipidaemia and medically treated hypertension
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders besides polyneuropathy
* Chronic or relevant acute infections (e.g. HIV, Hepatitis)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial except allowed co-medication
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 40 g/day = 5 units/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range and the clinical relevance is not acceptable (or the value is more than three times higher than the upper limit of the normal range e.g. liver enzymes)
* Change of drug dosing of allowed co-medication (anti-hypertensive agents, acetylic salicylic acid and statins) within the last 3 months
* Fasted blood glucose > 240 mg/dl (=13.3 mmol/L) on two consecutive days during washout
* Serum creatinine above upper limit of normal at screening

Male Patients:

* Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until one month after the last intake

Female patients:

* Positive pregnancy test

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Assessment of tolerability by investigator on a 4-point scale | Day 50
Incidence of adverse events | up to 50 days
Number of patients with abnormal changes in clinical laboratory parameters | Baseline, up to day 50

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | before and up to 43 days after first study drug administration
tmax (time from dosing to maximum concentration) | before and up to 43 days after first study drug administration
AUC (area under the concentration-time curve of the analyte in plasma) for several time points | before and up to 43 days after first study drug administration
Cmax,ss (maximum concentration of the analyte in plasma at steady state over a uniform dosing interval) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
Cpre,N (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N) | pre-dose on day 28
tmax,ss (time from dosing to maximum concentration at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
AUCτ,ss (area under the concentration time curve of the analyte in plasma at steady state over a uniform dosing interval) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
λz,ss (terminal rate constant in plasma at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
MRTpo,ss (mean residence time of the analyte in the body after 12 administrations at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
PTF (peak trough fluctuation) | before and 0:30 h, 1 h, 1:30 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 12 hours after last study drug administration
Accumulation ratio (RA) based on Cmax | up to 28 days
RA,AUC based on AUCτ | up to 28 days
Dipeptidyl-Peptidase IV (DPP-IV) activity for several time points | up to day 43
Change in fasting plasma glucose (AUEC0-3) after MTT (meal tolerance test ) | days -1, 1 and 29
Plasma glucose levels | up to day 43